CLINICAL TRIAL: NCT04133051
Title: Perioperative Analgesic Efficiency of Ultrasound Guided Quadratus Lumborum Block Versus Epidural Analgesia in Bladder Cancer Patients Undergoing Radical Cystectomy
Brief Title: Perioperative Analgesic Efficiency of Quadratus Lumborum Block vs Epidural in Radical Cystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AP1811-30103
Record Dates: First submitted 2019-08-12; First posted 2019-10-21 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative
Keywords: quadratus lumborum block; epidural analgesia; bladder cancer; radical cystectomy
MeSH Terms: conditions — Pain, Postoperative; Urinary Bladder Neoplasms | interventions — Tea

STUDY DESIGN:
Intervention Model Description: Group (A): 17 cases will be subjected to bilateral Ultrasound-guided Quadratus lumborum block through bilateral catheter insertion for perioperative analgesia.
  Group (B): 17 cases will be subjected to epidural catheter insertion for perioperative analgesia (as a control group).
  This number is to be increased to 34 patients (17 patients in each group) to account for the necessity to use non-parametric test. Sample size was calculated using G*Power program (University of Düsseldorf, Düsseldorf, Germany) 17, 20, 21.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Active Comparator): 17 cases will be subjected to bilateral Ultrasound-guided Quadratus lumborum block through bilateral catheter insertion for perioperative analgesia.
  Interventions: Drug: Quadratus Lumborum Block Using Bupivacaine 0.2%
- Epidural Analgesia (Active Comparator): 17 cases will be subjected to epidural catheter insertion for perioperative analgesia (as a control group).
  Interventions: Drug: Epidural Analgesia Using Bupivacaine 0.25%

INTERVENTIONS:
Drug: Quadratus Lumborum Block Using Bupivacaine 0.2% — Ultrasound guided transmuscular approach for quadratus lumborum block using an 18 gauge Touhy's epidural needle to insert the catheter. Normal saline 5 mL will be used to identify that plane. A volume of 20 ml of 0.25% of Bupivacaine bolus will be injected in that plane just over QL. This will be followed by epidural catheter insertion to facilitate continuous infusion. A similar procedure will be performed on the other side. A continuous infusion of 0.2% Bupivacaine at 5 ml/h will be administered to the patient.
  This transmuscular quadratus lumborum (TQL) block, has been suggested to be a simple and perhaps safer alternative to the anterior approach as was described for the original QL block
  Other Names: Transmuscular QL
  Arms: Quadratus Lumborum Block
Drug: Epidural Analgesia Using Bupivacaine 0.25% — With Patients placed in sitting position, puncture site will be identified at (T8-9, T9-10, or T10-11) intervertebral spaces. Using aseptic conditions, an 18G Tuohy epidural needle will be used to insert epidural catheter as appropriate.
  Induction of epidural analgesia with 10-15 ml bupivacaine 0.25% preoperatively with top up doses of 5-7 ml bupivacaine 0.25% or equivalent administered judiciously till we achieve analgesic level of T4 to L1. The calculated top up doses will be administered each hour using bupivacaine 0.25% or by using a continuous infusion syringe pump for equivalent doses
  Other Names: Thoracic Epidural
  Arms: Epidural Analgesia

SUMMARY:
This study is performed to measure the perioperative analgesic efficiency of bilateral quadratus lumborum block versus epidural analgesia in bladder cancer patients undergoing radical cystectomy

DETAILED DESCRIPTION:
1. Background and rationale:

   Bladder cancer is the ninth most common cancer in the world while being considerably common in both developed and developing countries. Bladder cancer is the most common malignancy among Egyptian males and it had been previously attributed to Schistosoma infection, a major risk factor for squamous cell carcinoma (SCC). Recently, transitional cell carcinoma (TCC) incidence has been increasing while SCC has declined. Exposures to tobacco smoke, occupational toxins, and environmental sources of heavy metals such as arsenic are the major reported risk factors for TCC .

   Acute perioperative pain management has been a matter of attention especially in major abdominal surgeries like radical cystectomy. Poor perioperative pain management especially with major abdominal surgeries can lead to deterioration of both physiological and psychological status of the patient leading to anxiety, stress, and patient's dissatisfaction while also leading to severe abdominal pain and diminished respiratory functions due to impaired function of accessory respiratory muscles which may precipitate shallow breathing, atelectasis, retained secretions, and also lack of patient's cooperation.

   Adequate multimodal perioperative pain management improves patient's recovery and survival on a general prospective due to decreased surgical stress response leading to better immunological functions and coagulation profile, and hence improving the outcome of the surgery.

   Perioperative epidural analgesia has been associated with improved overall survival but not reduced cancer recurrence. However, patients receiving epidural analgesia with or without general anesthesia have shown longer survival over 5 years period postoperatively than those receiving general anesthesia alone which can be related to better immunological profile and decreased stress response in regional anesthesia group of patients.

   Epidural analgesia for perioperative pain management has proven earlier recovery in post anesthesia care unit (PACU) with better pain and respiratory tolerance and decreased need for intravenous opioid administration. Perioperative continuous epidural analgesia was found to reduce hospital stay for patients undergoing major abdominal surgeries.

   Quadratus lumborum (QL) block was first described by Blanco and was previously called (the posterior approach of TAP block). Volunteers for QL spread of local anesthetic have shown a good spread of local anesthetics from T4 to L1 proving adequacy of QL block for analgesia over both posterior and anterior abdominal region surgeries. Further studies are being made to assess the adequacy of QL block as an analgesic technique for major abdominal surgeries.

   Perioperative analgesia using QL block with the ipsilateral technique following minor abdominal surgeries has shown decreased need for intravenous administration of opioids and has also shown promising results for adequate perioperative analgesia after major abdominal surgeries.

   Many reports have suggested that QL block can provide adequate analgesia not only for abdominal wall somatic pain but for severe visceral pain as well. The mechanism for visceral pain analgesia is not fully understood but it is suggested to be due to paravertebral spread of the injected local anesthetic.

   Early post-operative ambulation of bladder cancer patients undergoing radical cystectomy can be achieved using QL block which have a positive impact on both surgical outcome and patient survival. Radical cystectomy patients receiving QL block have shown decreased hospital stay with earlier discharge due to adequate long lasting analgesia and early ambulation.
2. Objectives:

   Primary Outcome:

   To test feasibility, efficiency, and safety of continuous perioperative QL block for perioperative pain management in bladder cancer patients undergoing radical cystectomy in comparison to continuous perioperative epidural analgesia for the same surgical procedure.
3. Study Design:

   * This study will be Prospective Randomized Controlled Study.
   * The study will be submitted to the Institutional Review Board (IRB) for review.
4. List of Correlative Studies:

   * Blanco R, Ansari T, Girgis E (2015): Quadratus lumborum block for postoperative pain after caesarean section: a randomised controlled trial. European Journal of Anaesthesiology (EJA). 32(11):812-8.
   * Blanco R, Ansari T, Riad W, & Shetty N (2016). Quadratus lumborum block versus transversus abdominis plane block for postoperative pain after cesarean delivery: a randomized controlled trial. Regional anesthesia and pain medicine, 41(6), 757-762.
5. Study Methods:

   • Interventions:

   Pre-interventional preparation:
   * Sedation for all patients prior to analgesic procedure at preoperative preparatory room using midazolam (0.02 mg/kg) intravenously.
   * Patients will be re-instructed about our anesthetic procedure steps according to each group.
   * Standard ASA monitoring for all patients before and during the anesthetic procedure.
   * Anesthetic procedure will start at the preoperative preparatory room in the form of regional block according to each of the study groups with catheter insertion and assessment of procedure success as discussed later.
   * Patients will be subjected to either quadratus lumborum block or epidural catheter insertion and analgesia as described later on.
   * Success of catheter insertion will be evaluated using 5ml of lidocaine 5% per catheter injection before proceeding with regular anesthetic doses. Analgesia level of T4 will be satisfactory for permitting transfer of patients to OR to proceed with general anesthesia and surgical procedure.
   * Routine assessment of all patients including assessment of patient's medical history, clinical examination, laboratory investigations (kidney and liver functions, CBC, and coagulation profile), ECG will be conducted on all patients above 40 years old and echocardiography for patients with suspected cardiomyopathies by medical history or preoperative examination. Chest X-ray for all patients suspected for respiratory diseases.
   * Patients will be subjected to continuous monitoring during surgery for any further complications related to anesthetic techniques and to surgery itself.
   * Patients will be monitored at PACU post-operatively to ensure hemodynamic stability, adequate analgesia, and attention for any possible complications that may occur due to anesthetic or surgical techniques used.
   * Patients will be discharged using the modified Aldrete's scoring system, a score of 9 or more will be sufficient for safe discharge of the patient to ward for further monitoring, continuation of analgesic techniques, and assessment of adequacy of analgesia post-operatively.
   * Patients' discharge time till reaching sufficient Aldrete's score for each study group will be calculated and included in the study parameters for further assessment of safety and efficiency of analgesic techniques used.

     • Possible risks:
   * Orthostatic hypotension.
   * Hemodynamic instability (e.g. bradycardia, ECG changes, tachycardia).
   * Local anesthetic toxicity.

     * Source of Funding:

   No source of funding.
   * Time plan:

     * The study is to be started in 2018 and is expected to be finished in 2020.
     * The expected publishing date is 2020.
   * Benefits from the study:

   To test feasibility, efficiency, and safety of continuous perioperative QL block for perioperative pain management in bladder cancer patients undergoing radical cystectomy in comparison to continuous perioperative epidural analgesia for the same surgical procedure.

   • Possible Risk:
   * Orthostatic hypotension.
   * Hemodynamic instability (e.g. bradycardia, ECG changes, tachycardia).
   * Local anesthetic toxicity.
6. Protection of privacy and confidentiality of patients' information:

   Data collection and presentation will be anonymous and both privacy and confidentiality will be protected to the maximal possible standards.
7. Publication policy:

Any article arising from this work will carry the names of all participants with the name orders according to the degree of contribution to data interpretation and manuscript writing. Additional external authors may be added if they add to the content and qualify for authorship by the international standards.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III
* Adult patients (>18 years old)
* Both sexes
* Scheduled for radical cystectomy at NCI, CU

Exclusion Criteria:

* Patient's refusal of the study procedures
* Allergy to drugs used in the study
* Patients with chronic pain
* Patients with coagulopathies (INR > 1.6 or platelets count < 50,000 cc3)
* Hemodynamically unstable patients (e.g. BP < 90/60)
* Patients with local or intra-abdominal infections concerning intervention sites and septic patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain (VAS) score measurement postoperatively | 0 Hours Postoperatively
  The primary outcome measures visual analogue pain scores in the two groups at the end of surgery
Visual analogue pain (VAS) score measurement 6 hours postoperatively | 6 Hours Postoperatively
  The primary outcome measures visual analogue pain scores in the two groups 6 hours postoperatively
Visual analogue pain (VAS) score measurement 24 hours postoperatively | 24 Hours Postoperatively
  The primary outcome measures visual analogue pain scores in the two groups 24 hours postoperatively
Visual analogue pain (VAS) score measurement 48 hours postoperatively | 48 Hours Postoperatively
  The primary outcome measures visual analogue pain scores in the two groups 48 hours postoperatively

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting | 48 Hours Postoperatively
  Postoperative Nausea and Vomiting using nausea score (0 for none, 1 for mild to moderate nausea, 2 for moderate nausea, 3 for severe nausea accompanied by vomiting) When patient's nausea score reaches ≥ 2; intravenous anti-emetics in the form of Ondasetron 8mg and will be administered and recorded in all groups

OTHER OUTCOMES:
Morphine Usage | 48 Hours Postoperatively
  During pain assessment using visual analogue score, if VAS score is ≥ 4, intravenous morphine 3mg will be administered 18. The mean first time for morphine requirement will be recorded in all groups (mean+- SD). Total 48 h morphine consumption will be recorded in all groups
Patient's satisfaction | 48 Hours Postoperatively
  Patient satisfaction with the technique and analgesia to be assessed at the end of study (at 48 hours period) and will be put on a scale from 1 to 4 (poor = 1, fair = 2, good = 3, excellent = 4)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H. Bakeer, M.D., Study Director — National Cancer Institute, Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488